CLINICAL TRIAL: NCT05420623
Title: Determination and Evolution of Usual Locomotion Strategies of Lower Limb Amputees by Gait Analysis
Brief Title: Walking Strategies in Usual Locomotion of Lower Limb Amputees
Acronym: STRAAL
Status: Completed | Type: Observational
Sponsor: FondationbHopale (Other)
Collaborators: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: HOP-RIPH2-21-01
Record Dates: First submitted 2021-12-13; First posted 2022-06-15 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2023-08

CONDITIONS: Lower Limb Amputation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Amputees patients
- control group: non-amputees

SUMMARY:
Amputation is a life-altering event with an immediate and obvious effect on daily life activities and quality of life. Asymmetrical movements of the lower limbs and compensatory strategies during walking are associated with an elevated risk for developing deleterious secondary health conditions. It is well established that therapeutic gait training methods are effective in reducing spatiotemporal gait deviations and improving functional mobility. However, the littérature does not clearly indicate the best time to perform a gait training or which gait parameters predict it.

The main aim of this study is to determinate the walking strategies of lower limb amputees in several locomotion tasks on daily life. Then, the investigators study the evolution of these walking strategies after a gait training and over time.

DETAILED DESCRIPTION:
Quantified gait analyses are included in the practice for consultations to monitor orthopaedic devices, and are specific to the study for the rehabilitation stay (V2 and V3).

The subjects in the control group will be recruited from among the carers of patients undergoing rehabilitation and from among volunteers recruited by means of posters in the establishments of the HOPALE Foundation in Berck.

Once the eligibility criteria have been checked, a quantified gait analysis and functional tests will be carried out: the 6-minute walk test (T6M) and the Time Up and Go test (TUG). They will complete a single visit lasting approximately 1 hour and 30 minutes.

ELIGIBILITY:
Inclusion Criteria (Amputees patients):

* Major amputation of the lower limb,
* Unilateral amputation,
* Aged 18 or over,
* Mobility level equal to or greater than 2 (according to Medicare Functional Classification Levels),
* Subject who has given his or her free and informed consent.

Non-inclusion Criteria (Amputees patients):

* Definitive apparatus less than one month old,
* Contraindications for walking,
* Presence of a major neurocognitive disorder reported in the medical record (as mentioned in the DMS-5): acquired, significant and progressive reduction in abilities in one or more cognitive domains, significant enough to no longer be able to perform activities of daily living alone (loss of autonomy)
* Cognitive disorders reported in the medical file,
* Subject under guardianship, curatorship or protective measure,
* Pregnant or lactating woman.

Inclusion Criteria (Healthy volunteers):

- Able to walk 50m alone.

Non- Inclusion Criteria (Healthy volunteers):

* Contraindication to effort,
* Cognitive disorders known by the subject, causing difficulties in performing tasks related to activities of daily living
* Any history of neurological or orthopedic origin likely to limit the quality of walking,
* Notion of trauma on the musculoskeletal system less than 3 months (sprain type, muscle injury, etc.),
* Subject under guardianship, curatorship or protective measure,
* Pregnant or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Visits are carried out as part of routine care, either in the case of a follow-up consultation, or as part of a scheduled entry into a rehabilitation center.
  If the patient is included at the entrance of a scheduled rehabilitation stay, the data from his last follow-up consultation will be recovered retrospectively (follow-up AQM + functional tests).
  Recruitment of healthy volunteers :
  The study will be offered to the companions of people followed in rehabilitation at the Jacques Calvé center. Posters will be placed at the reception desk of the institution and in the consultation waiting rooms.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Data from the quantified gait assessment: walking speed (m/s) | Inclusion
  Full body motion capture was systematically analyzed for different walking conditions
  * normal and fast walking on self selected walking speed, walking on cross-slope, go up and down a step, and turn.
Data from the quantified gait assessment: step length (m) | Inclusion
  Full body motion capture was systematically analyzed for different walking conditions
  * normal and fast walking on self selected walking speed, walking on cross-slope, go up and down a step, and turn.
Data from the quantified gait assessment: step time (s) | Inclusion
  Full body motion capture was systematically analyzed for different walking conditions
  * normal and fast walking on self selected walking speed, walking on cross-slope, go up and down a step, and turn.
Data from the quantified gait assessment: lower limbs joint angles (degrees) | Inclusion
  Full body motion capture was systematically analyzed for different walking conditions
  * normal and fast walking on self selected walking speed, walking on cross-slope, go up and down a step, and turn.
Data from the quantified gait assessment: joint moments (N.m/kg) | Inclusion
  Full body motion capture was systematically analyzed for different walking conditions
  * normal and fast walking on self selected walking speed, walking on cross-slope, go up and down a step, and turn.
Data from the quantified gait assessment: trunk and pelvis position (degrees) | Inclusion
  Full body motion capture was systematically analyzed for different walking conditions
  * normal and fast walking on self selected walking speed, walking on cross-slope, go up and down a step, and turn.
Data from the quantified gait assessment: ground reaction forces (N). | Inclusion
  Full body motion capture was systematically analyzed for different walking conditions
  * normal and fast walking on self selected walking speed, walking on cross-slope, go up and down a step, and turn.

SECONDARY OUTCOMES:
The correlations between some data from clinical assessment and gait parameters are analyzed : pain scale (Numerical Rating Scale) | Inclusion
The correlations between some data from clinical assessment and gait parameters are analyzed : strenght testing of hip abductor/extensor/flexor and knee extensor/flexor (if applicable) | Inclusion
  This measurement will be collected with handheld dynamometer (Newton)
The correlations between some data from clinical assessment and gait parameters are analyzed : amputation level and etiology, prosthesis characteristics, lower limbs range of motion with manual goniometer (degrees) | Inclusion
The correlations between some data from clinical assessment and gait parameters are analyzed : amputation level and etiology, prosthesis characteristics, functional walking tests (timed up and go test - in seconds). | Inclusion
The correlations between some data from clinical assessment and gait parameters are analyzed : amputation level and etiology, prosthesis characteristics, functional walking tests (six minute walk test - in meters). | Inclusion
These clinical assessment and these gait parameters on the conditions mentioned are analyzed before and after rehabilitation during consultations, and then at 6 months and at 12 months : pain scale (Numerical Rating Scale) | Inclusion, 6 months, 12 months
These clinical assessment and these gait parameters on the conditions mentioned are analyzed before and after rehabilitation, and at 6 and 12 months: strenght testing of hip abductor/extensor/flexor and knee extensor/flexor (if applicable) | Inclusion, 6 months, 12 months
  This measurement will be collected with handheld dynamometer (Newton)
These clinical assessment and these gait parameters on the conditions mentioned are analyzed before and after rehabilitation during consultations, and then at 6 months and at 12 months : lower limbs range of motion with manual goniometer (degrees) | Inclusion, 6 months, 12 months
These clinical assessment and these gait parameters on the conditions mentioned are analyzed before and after rehabilitation during consultations, and then at 6 months and at 12 months : functional walking tests (timed up and go test, in seconds) | Inclusion, 6 months, 12 months
The correlations between some data from clinical assessment and gait parameters are analyzed : amputation level and etiology, prosthesis characteristics, functional walking tests (six-minute walk test, in meters). | Inclusion, 6 months, 12 months
If you need a walking aid, the investigators compares the force applied to the walking aid, using a force sensor (Newton), with biomechanical compensations. | Inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Frederic CHARLATE, Principal Investigator — Fondation Hopale
Locations (1):
- Fondation HOPALE - Centre de rééducation Jacques CALVE, Berck, Hauts-de-France, France